CLINICAL TRIAL: NCT05499689
Title: Comparison of Transcutaneous Pulsed Radiofrequency Therapy and Greater Occipital Nerve Block Efficiency in Migraine Headache
Brief Title: Transcutaneous Pulsed Radiofrequency in Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Director, medical doctor, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Transcutaneous GON
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Migraine Disorders
Keywords: Transcutaneous pulsed radiofrequency; pulsed radiofrequency treatment; headache; GON block
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GON block group (Active Comparator): 30 patients who underwent greater occipital nerve block
  Interventions: Drug: Bupivacaine Hydrochloride
- Transcutaneous pulsed RF group (Active Comparator): 30 patients who underwent greater occipital nerve pulsed radiofrequency
  Interventions: Other: Transcutaneous pulsed radiofrequency qurrent

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — 2.5 cc bupivacain injection will be administered by approaching the greater occipital nerve under ultrasound guidance.
  Arms: GON block group
Other: Transcutaneous pulsed radiofrequency qurrent — Pulsed radiofrequency current will be applied through transcutaneous pads adhered over the greater occipital nerve trace on the nape.
  Arms: Transcutaneous pulsed RF group

SUMMARY:
The aim of the investigator is to compare the efficacy of greater occipital nerve block and transcutaneous pulsed radiofrequency treatment in migraine.

DETAILED DESCRIPTION:
Migraine is the second most common primary headache. Greater occipital nerve (GON) block is an effective method in the treatment of migraine. Transcutaneous pulsed radiofrequency (RF) therapy is used in the treatment of pain. However, its use in headaches is not widespread yet.

Investigator aimed to compare the efficacy of transcutaneous pulsed radiofrequency therapy applied through the GON trace and GON block therapy. A 60-patient study was designed. GON block was planned for 30 patients and transcutaneous pulsed RF was planned for 30 patients. The block will be applied once at the level of C2 vertebra with ultrasound.Transcutaneous pulsed RF will be applied twice, once a week, for 8 minutes.All patients will have pre-treatment migraine disability assessment score (MIDAS) scores filled. A headache diary will be provided to all patients. Frequency and severity of pain will be followed for 1 month. Pain intensity will be evaluated on the visual analog scale (VAS).

Investigator aimed to evaluate the efficacy of transcutaneous pulsed RF therapy, which is a noninvasive method, in migraine.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Migraine

Exclusion Criteria:

* Other headaches will not accompany (tension-type headache, cluster...)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2023-06-22 (Estimated); Study Completion 2023-08-22 (Estimated)

PRIMARY OUTCOMES:
The Migraine Disability Assessment Test | Baseline
  The MIDAS questionnaire is an important part of a package of educational, investigative, and therapeutic measures, and could play a major role in improving the care of patients with migraine and other types of headache.

SECONDARY OUTCOMES:
Visual analog scale (VAS) | Baseline, Week 4
  It is a scale that measures the severity of pain. Scored between ''0: no pain'' and ''10: worst pain'' .

CONTACTS AND LOCATIONS:
Overall Officials: mehlika panpallı ateş, Study Chair — Diskapi TRH; ömer taylan akkaya, Study Director — Diskapi TRH; Hüseyin Alp Alptekin, Study Chair — Diskapi TRH
Locations (1):
- Diskapi Yildirim Beyazıt Teaching and Research Hospital, Ankara, Altındğ, Turkey (Türkiye)

REFERENCES:
- [Derived] Perdecioglu GRG, Ates MP, Yuruk D, Can E, Yildiz G, Akkaya OT. A new neuromodulation method in chronic migraine; non-invasive pulsed radiofrequency, a single-blinded, randomised, controlled trial. Ir J Med Sci. 2024 Jun;193(3):1487-1493. doi: 10.1007/s11845-023-03598-x. Epub 2023 Dec 26. PMID 38147268